CLINICAL TRIAL: NCT05106621
Title: NEW MODEL OF ORGANIZATION OF AN OPERATIVE BLOCK (BLOC-OP)
Brief Title: AN INTELLIGENT MODEL FOR THE OPERATIVE BLOCK
Acronym: BLOC-OP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Chief of 2^ UO Anesthesua and Intensive Care, Full Professor of University of Parma, University of Parma
Other Study IDs: 1284/2020/OSS/AOUPR
Record Dates: First submitted 2021-10-11; First posted 2021-11-04 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Artificial Intelligence in Operating Room
Keywords: Perioperative Medicine; Artificial Intelligence; Machine Learning; Operating Room

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Patients

SUMMARY:
Perioperative medicine is characterized by a very delicate path; it is composed, in fact, of a series of highly specialized clinical measures managed by various professionals (surgeons, anesthetists, intensivists, nurses, etc.), who work together to ensure the best quality of all phases of the path (preoperative , intra and postoperative). On the other hand, it is necessary to underline the huge resources needed to provide surgical services. Organizational optimization, based on specific analyzes, could lead to a more careful management of resources in this area, avoiding waste due to early closure of the operating room or unexpected extension of the same. In recent years, precisely to respond to the need to analyze large quantities of information, the use of artificial intelligence techniques, and in particular of machine learning, is becoming increasingly popular, a branch of artificial intelligence that aims, through the use of algorithms and statistical model, to infer new knowledge in a way automatic. Such technologies appear to possess excellent analytical skills both in the clinical and, above all, organizational fields. The data that are emerging in the literature on this issue, although still the first in this regard, seem to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

all patients undergoing surgery who sign the informed consent form will be included.

Exclusion Criteria:

refusal of the patient to the study in question.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing abdominal, thoracic, urological, vascular, orthopedic and gynecological and plastic surgery
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Time Prediction | 1 year
  Prediction of time spend in oprating room

SECONDARY OUTCOMES:
Outcome evaluation | 1 year
  ICU admission
Outcome evaluation | 1 year
  Rate of surgical procedures cancellation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera-Universitaria di Parma, Parma, Italy

REFERENCES:
- [Background] Evans RS, Burke JP, Classen DC, Gardner RM, Menlove RL, Goodrich KM, Stevens LE, Pestotnik SL. Computerized identification of patients at high risk for hospital-acquired infection. Am J Infect Control. 1992 Feb;20(1):4-10. doi: 10.1016/s0196-6553(05)80117-8. PMID 1554148
- [Background] Redfern RO, Langlotz CP, Abbuhl SB, Polansky M, Horii SC, Kundel HL. The effect of PACS on the time required for technologists to produce radiographic images in the emergency department radiology suite. J Digit Imaging. 2002 Sep;15(3):153-60. doi: 10.1007/s10278-002-0024-5. Epub 2002 Nov 6. PMID 12415466
- [Background] Lee TT, Liu CY, Kuo YH, Mills ME, Fong JG, Hung C. Application of data mining to the identification of critical factors in patient falls using a web-based reporting system. Int J Med Inform. 2011 Feb;80(2):141-50. doi: 10.1016/j.ijmedinf.2010.10.009. Epub 2010 Nov 5. PMID 21115393
- [Background] Martins M. Use of comorbidity measures to predict the risk of death in Brazilian in-patients. Rev Saude Publica. 2010 Jun;44(3):448-56. doi: 10.1590/s0034-89102010005000003. Epub 2010 Apr 30. PMID 20428601
- [Background] Izad Shenas SA, Raahemi B, Hossein Tekieh M, Kuziemsky C. Identifying high-cost patients using data mining techniques and a small set of non-trivial attributes. Comput Biol Med. 2014 Oct;53:9-18. doi: 10.1016/j.compbiomed.2014.07.005. Epub 2014 Jul 22. PMID 25105749
- [Derived] Bottani E, Bellini V, Mordonini M, Pellegrino M, Lombardo G, Franchi B, Craca M, Bignami E. Internet of Things and New Technologies for Tracking Perioperative Patients With an Innovative Model for Operating Room Scheduling: Protocol for a Development and Feasibility Study. JMIR Res Protoc. 2023 Jul 5;12:e45477. doi: 10.2196/45477. PMID 37405821